CLINICAL TRIAL: NCT04025450
Title: Comparation of Chidamide Plus VRD (Bortezomib, Lenalidomide, Dexamethasone) With VRD Regimen for Primary High-Risk Multiple Myeloma Patients, a Phase I/II, Multiple Center, Randomized Clinical Trial
Brief Title: Comparation of Chidamide Plus VRD (Bortezomib, Lenalidomide, Dexamethasone) With VRD Regimen for Primary High-Risk Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ChiVRD VS VRD-MM02
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: In this trial, patients will be randomly assigned to chidamide+VRD group or VRD group, and then treated with the corresponding regimen, and their safety and efficacy will be evaluated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide plus VRD (Experimental): Chidamide:30mg d0,d3,d7,d10/Velcade:1.3mg/m2 d1,d4,d8,d11/ Dexamethasone: 10mg BID d1,d2,d4,d5,d8,d9,d10,d11/Lenalidomide: 25mg d1-d14
  Interventions: Drug: Chidamide+VRD
- VRD (Active Comparator): Velcade:1.3mg/m2 d1,d4,d8,d11/ Dexamethasone: 10mg BID d1,d2,d4,d5,d8,d9,d10,d11/Lenalidomide: 25mg d1-d14
  Interventions: Drug: VRD

INTERVENTIONS:
Drug: Chidamide+VRD — Chidamide:30mg d0,d3,d7,d10/Velcade:1.3mg/m2 d1,d4,d8,d11/ Dexamethasone: 10mg BID d1,d2,d4,d5,d8,d9,d10,d11/Lenalidomide: 25mg d1-d14
  Arms: Chidamide plus VRD
Drug: VRD — Velcade:1.3mg/m2 d1,d4,d8,d11/ Dexamethasone: 10mg BID d1,d2,d4,d5,d8,d9,d10,d11/Lenalidomide: 25mg d1-d14
  Arms: VRD

SUMMARY:
In the phase I trial, dose escalation of chidamide will be performed at 4 different dosages (15mg, 20mg, 25mg, 30mg) for optimal dosage, in the phase II trial, the safety and efficacy of chidamide+VRD will be compared with that of VRD regimen.

DETAILED DESCRIPTION:
In the phase I trial, dose escalation of chidamide will be performed at 4 different dosages (15mg, 20mg, 25mg, 30mg) for optimal dosage, which will be determined by efficacy and safety profiles of the patients; afterward, the optimal dosage of chidamide will be combined with VRD regimen, patients will be randomly assigned to chidamide+VRD group or VRD group, and their efficacy and safety will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed as multiple myeloma, and has one of the above:

  1. high risk karyotype, such as 17p-，t（4；14），t（14；16），t（14；20）或1q gain,1p-, double hit myeloma, triple hit myeloma, etc;
  2. RISS-3;
  3. IgD/IgE MM;
  4. with measurable extra-medullary plasmacytoma;
  5. flowcytometry showed peripheral blood plasma cell ≥0.165%；
* 2.Secretory MM should have measurable markers, including:

  1. specific M protein value (≥5g/L)；
  2. and/or involved flc ≥100mg/L；
  3. and/or measurable extramedullary foci (diameter>1cm on CT);
* 3.Age≥18 years, male or female;
* 4.ECOG 0-2 points, with life expectance ≥3 months; GA score <2;
* 5.ALT/AST level <2.5 times of the maximum of normal range; total bilirubin<1.5 times of normal maximum；
* 6.Neutrophil count≥1.5×109/L, platelet count≥50×109/L;
* 7.eGFR≥40ml/min，except in the case of myeloma-related nephropathy;
* 8.Normal left ventricular ejaculation rate, NYHA stage 1, pulmonary function GOLD stage 1;
* 9.Willing to accept the possibility of potential adverse events and efficacy observation by the investigators;
* 10.Being able to understand and signing the written consent, which should be signed prior to any procedure of the trial.

Exclusion Criteria:

* 1.With ≥2 degree of peripheral neuropath or with pain;
* 2.Having received any of the medicine of the experiment regimen within 30 days prior to enrollment, pain-relieving radiotherapy is allowed;
* 3.With severe pulmonary/cardiac disfunction (including history of QT interval elongation, ventricular tachycardia, ventricular fibrillation, myocardial infraction) or other severe organ malfunction;
* 4.Patients in pregnancy or lactation;
* 5.Allergic constitution or being allergic to any drug within the regimen of the trial;
* 6.With uncontrolled mental diseases;
* 7.With active infection;
* 8.With non-myeloma-associated acute renal dysfunction;
* 9.With active hepatitis;
* 10.HIV positive;
* 11.History of other malignant tumor within 5 years prior to enrollment; except for the case of in situ cervical cancer and non-malignant melanoma;
* 12.With other conditions that the investigators think unfit for the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | at the time point 1 month after the last cycle
  complete remission rate after treated by the corresponding regimen
incidence and severity of adverse events | from the date of the start of treatment to 36 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

SECONDARY OUTCOMES:
progression free survival | from the day of treatment to the date of first documented progression，up to 36 months after the last patient's enrollment;
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | from the day of treatment to the date of first documented progression，up to 36 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: chengcheng Fu, PhD, Principal Investigator — First Affiliated Hospital of Suzhou University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China